CLINICAL TRIAL: NCT03063008
Title: "Randomized Evaluation of Bone Ingrowth After Intervertebral Body Fusion With Either MectaLIF® PEEK or MectaLIF® TiPEEK Oblique"
Brief Title: Transforaminal Lumbar Interbody Fusion in PEEK Oblique Cages With and Without Titanium Coating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammad ARAB MOTLAGH (Other)
Responsible Party: Sponsor-Investigator, Mohammad ARAB MOTLAGH, MD, PhD, Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TiPEEK Cage
Record Dates: First submitted 2017-02-16; First posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Vertebral Fusion
Keywords: Lumbar spine; Fusion; Titanium; PEEK

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbar fusion with PEEK cage (Other): Control arm
  Interventions: Device: PEEK
- Lumbar fusion with TiPEEK cage (Other): Study arm
  Interventions: Device: TiPEEK

INTERVENTIONS:
Device: PEEK — Procedure/Surgery:
  TLIF fusion with common PEEK cages.
  Arms: Lumbar fusion with PEEK cage
Device: TiPEEK — Procedure/Surgery:
  TLIF fusion with titanium coated PEEK cages.
  Arms: Lumbar fusion with TiPEEK cage

SUMMARY:
Clinical outcome with regard to oswestry disability index and lumbar fusion rate after implantation of titanium coated PEEK cage and common PEEK cage

DETAILED DESCRIPTION:
Cages made of polyetheretherketone (PEEK) and titanium materials reliably produce successful fusion rates and good clinical outcomes. However, there is a paucity of studies that have assessed the optimal material of cage systems. The primary objective of this study was to compare the Oswestry Disability Index (ODI) after instrumented transforaminal lumbar interbody fusion (TLIF) using either titanium-coated polyetheretherketone (TiPEEK) or common PEEK cages. Secondary objectives were to assess differences in fusion rates and differences in pain and in quality of life between these groups.

ELIGIBILITY:
Inclusion Criteria:

Persistence of

* low back pain,
* sciatica and
* spinal claudication after conservative treatment attributed to L3 to L5 lumbar segments.

Exclusion Criteria:

* previous lumbar spinal surgery
* body mass index >35 kg/m²

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01-16 (Actual); Primary Completion 2013-09-01 (Actual); Study Completion 2013-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical outcome assessed by Oswestry Disability Index (ODI) after instrumented transforaminal lumbar fusion with TiPEEK or common PEEK | 12 months
  Oswestry Disability Index (ODI) after instrumented transforaminal lumbar fusion with TiPEEK or common PEEK

SECONDARY OUTCOMES:
Fusion result | 12 months
  Fusion rate after instrumented transforaminal lumbar fusion with TiPEEK or common PEEK

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Arabmotlagh, MD, PhD, Study Director — Department of Orthopedic Surgery, University Hospital Frankfurt

IPD SHARING:
Plan to Share IPD: No